CLINICAL TRIAL: NCT03200067
Title: Effects on the Personalized Rehabilitation Service in Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Eun Joo Yang, Study chair, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: B-1705/395-302
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Last update posted 2017-06-27 (Actual); Status verified 2017-06

CONDITIONS: Breast Cancer; Breast Neoplasms; Breast Cancer Female; Lymphedema
MeSH Terms: conditions — Breast Neoplasms; Lymphedema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized rehabilitation service group (Experimental): Breast cancer patients who use mobile healthcare service application and receive personal feedback from clinician
  Interventions: Behavioral: Personalized health care service
- Conventional group (No Intervention): Breast cancer patients with conventional care

INTERVENTIONS:
Behavioral: Personalized health care service — Personalized health care service, such as rehabilitation exercise recommendation, lifestyle activity coaching, health data monitoring
  Arms: Personalized rehabilitation service group

SUMMARY:
In order to study the effectiveness of personalized healthcare service program for breast cancer rehabilitation, investigators designed this study using mobile phone and clinical intervention(feedback coaching).

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patient (age over 18), Cancer stage under 3, Android OS smartphone user

Exclusion Criteria:

* Cancer stage over 4, Patients diagnosed with multiple cancer, Patient who cannot participate rehabilitation exercise program

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-06-03 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-09 (Estimated)

PRIMARY OUTCOMES:
Patient health ability change | Baseline and after 4 weeks, 8 weeks of lifestyle modification
  Measuring Health and Disability WHODAS 2.0

SECONDARY OUTCOMES:
Lab test result change | Baseline and after 4 weeks, 8 weeks of lifestyle modification
  Laboratory test (Blood test)
Patient satisfaction change on mobile service | Baseline and after 4 weeks, 8 weeks of lifestyle modification
  Patient subjective evaluation by survey on satisfaction
Patient satisfaction change on healthcare management | Baseline and after 4 weeks, 8 weeks of lifestyle modification
  Patient subjective evaluation by survey on satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Eunjoo Yang, PhD, Study Chair — Seoul National University Bundang Hospital
Locations (1):
- Seoul national university bundang hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No